CLINICAL TRIAL: NCT06683378
Title: Phase I Randomized, Double-blind Study to Evaluate Feasibility, Safety, and Clinical Responses of Implanting Autologous Peripheral Nerve Tissue Into the Nucleus Basalis of Meynert or Substantia Nigra for Non-motor or Motor Symptoms in Patients With Parkinson's Disease Undergoing DBS Surgery
Brief Title: A Study to Evaluate Feasibility, Safety, and Clinical Responses of Implanting Autologous Peripheral Nerve Tissue Into the Brain for Non-motor or Motor Symptoms in Patients With Parkinson's Disease Undergoing DBS Surgery
Acronym: STAR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Craig van Horne, MD, PhD (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Craig van Horne, MD, PhD, Department of Neurosurgery Chair, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 90066; 1R01AG081356-01A1 (NIH)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Deep Brain Stimulation; DBS; Cell and Tissue Based Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peripheral nerve tissue (PNT) deployment to the Substantia Nigra (Active Comparator)
  Interventions: Procedure: Reparative Autologous peripheral nerve tissue
- Peripheral nerve tissue (PNT) deployment to the nucleus basalis of Meynert (Active Comparator)
  Interventions: Procedure: Reparative Autologous peripheral nerve tissue

INTERVENTIONS:
Procedure: Reparative Autologous peripheral nerve tissue — At the time participants are receiving the standard of care deep brain stimulation (DBS) surgery, a standard incision on the lateral aspect near the ankle is made, the sural nerve is identified, an about 3 cm biopsy of the sural nerve is obtained and the incision is closed.
  From the biopsied section, the epineurium is removed, fascicles are cut, and (~5 pieces per side; ~ 5mm length x 1.5 mm diameter: approximately 10 cubic millimeters) implanted bilaterally into the nucleus basalis of Meynert (NBM) or substantia nigra (SN).

SUMMARY:
The investigators propose a Phase I single surgical-center, double-blinded randomized parallel clinical trial involving bilateral autologous peripheral nerve tissue (PNT) delivery into the NBM or the alternate target also affecting cognition in this population, the substantia nigra (SN), to address "repair cell" support of these areas. Twenty-four participants with idiopathic Parkinson's Disease (PD) who have selected, qualified and agreed to receive as standard of care deep brain stimulation (DBS) will be enrolled and randomly allocated to receive bilateral PNT deployment to either the NBM or SN at the time of DBS surgery. Participants will be allocated equally among both assignments over the course of three years (8 Year 1, 10 Year 2, 6 Year 3). Participants will be evaluated for neurocognitive, motoric function, activities of daily living, and quality of life at enrollment before surgery, two-weeks after surgery, and 6, 12, and 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing DBS
* Diagnosis of clinically established or clinically probably PD as defined by MDS criteria
* Age 45-75, inclusive
* Able to tolerate the surgical procedure
* Able to undergo all planned assessments
* Available access to the sural nerve

Exclusion Criteria:

* Any condition that would not make the subject a candidate for DBS
* Dementia diagnosis
* Previous PD surgery or intracranial surgery
* Unable to undergo an MRI
* An obstructed trajectory path to the substantia nigra and nucleus basalis of Meynert

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Successful deployment of bilateral peripheral nerve tissue (PNT) into the brain | Intraoperative
  Number of participants in each study arm who successfully receive bilateral PNT delivery.
Number of participants completing 12 month study visit | 12-month study visit
  Total number of participants to complete study visit by arm assignment
Study-related adverse events as assessed by MedDRA v27 | Enrollment to 24-month study visit
  Total number of study-related adverse events experienced by participants.
Study-related serious adverse events as assessed by MedDRA v.27 | Enrollment to 24-month study visit
  Total number of serious adverse events experienced by participants

SECONDARY OUTCOMES:
PNT deployment attempts | During surgery
  Number of deployment attempts required, per participant, to deliver bilateral PNT by group allocation
Mean change in Montreal Cognitive Assessment (MoCA) scores | Baseline 6, 12 and 24 months after surgery
  Mean change in MoCA scores for participants at study visits compared to baseline by group allocation. Assessment is scored from 0-30 with a score of 26 or better indicating normal cognition. A score less than 26 indicates a cognitive deficit.
Mean change in Neuropsychological assessment scores | Baseline, 12 and 24 months
  Participants complete a neuropsychological assessment battery that meets the Movement Disorder Society (MDS) guidelines for determining mild cognitive impairment/mild neurocognitive disorder. Domains include attention and working memory, executive functioning, memory (verbal and visual), language, and visuospatial skills. Participants' raw scores will be converted to standardized scores based on appropriate norms (e.g., age-based norms). Participants' 12 and 24-month re-evaluation will be compared to their baseline pre-surgical assessment to determine change from baseline on each measure. A change that exceeds 1.5 standard deviation from their baseline performance will be considered notable.
Change in Neuropsychological diagnosis | Baseline, 12 and 24 months
  Changes in participant neuropsychological diagnoses during scheduled evaluations will be reported. e.g. No cognitive diagnosis progressing to mild neurocognitive disorder.
Change in Neuropsychological domains with impairment | At 12, 24 months compared to baseline
  A count of the number of domains with impairment at each study visit to compare with previous study visits.
Mean change in Modified Schwab and England Scale of Activities of Daily Living scores | At 6, 12, 24 months compared to baseline
  Mean change participant independence levels as measured in Schwab and England Scale of Activities of Daily Living scores. 100% = completed independent and 0% being completely dependent.
Mean change in Parkinson's Disease Questionnaire-8 (PDQ-8) quality of life scores | At 12 and 24 months compared to baseline
  Assess changes in participant's quality of life. Questionnaire is scored from 0-32 with higher scores indicating poorer quality of life.
Mean change in Non-motor symptom scale scores | At 12 and 24 months compared to baseline
  Assessment used to identify Parkinson's disease related non-motor symptoms experienced by participants. The scale measures the frequency and severity of symptoms and is scored from 0-360 with higher scores indicating more frequent and severe symptoms.
Mean change of the Movement Disorder Society - Unified Parkinsons Disease Rating Scale (MDS-UPDRS) Part I scores | 6, 12, and 24 months as compared to baseline
  MDS-UPDRS Part I scores non-motor symptoms effecting activities of daily living in those with Parkinson's Disease. Scores range from 0-52 with higher scores indicating greater symptom severity.
Mean change of the MDS-UPDRS Part II scores | At 6, 12, 24 months compared to baseline
  MDS-UPDRS Part II scores motor symptoms effecting activities of daily living in those with Parkinson's Disease. Scores range from 0-52 with higher scores indicating greater symptom severity.
Mean change in MDS-UPDRS Part III scores | At 6, 12, 24 months compared to baseline
  MDS-UPDRS Part III scores motor symptoms associated with Parkinson's Disease. Part III scores range from 0-132 with higher scores indicating higher symptom severity.
Mean change in MDS-UPDRS Part IV scores | At 6, 12, and 24 months compared to baseline
  MDS-UPDRS Part IV scores motor complications such as fluctuations and dyskinesia's associated with anti-Parkinson's medications. Scores range from 0-24 with higher scores indicating greater severity in motor complications.
Number of participants completing 24-month study visit | 24-month study visit
  Total number of participants completing 24 month study visit by group allocation
Mean change in Dementia Rating Scale (DSRS) | Baseline 6, 12 and 24 months after surgery
  A survey to assess and rate changes the cognitive and behavioral functioning of participants. Scale is scored from 0-54 with being higher numbers indicating greater dementia severity.

CONTACTS AND LOCATIONS:
Overall Officials: Craig G van Horne, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
The focus of this study is PD, but images and results will be made available to other researchers by asking participants, at the time of consent, their willingness to permit sharing of data and bio-specimens.

REFERENCES:
- [Background] Quintero JE, Chau MJ, Slevin JT, Koehl L, Gurwell JA, Wallace E, Kryscio RJ, El Khouli R, Anderson-Mooney AJ, Schmitt FA, Gerhardt GA, van Horne CG. Two-year feasibility and safety of open-label autologous peripheral nerve tissue implantation during deep brain stimulation in patients with Parkinson's disease. J Parkinsons Dis. 2025 Mar;15(2):397-408. doi: 10.1177/1877718X241312409. Epub 2025 Feb 25. PMID 40007169
- [Background] van Horne CG, Quintero JE, Slevin JT, Anderson-Mooney A, Gurwell JA, Welleford AS, Lamm JR, Wagner RP, Gerhardt GA. Peripheral nerve grafts implanted into the substantia nigra in patients with Parkinson's disease during deep brain stimulation surgery: 1-year follow-up study of safety, feasibility, and clinical outcome. J Neurosurg. 2018 Dec 1;129(6):1550-1561. doi: 10.3171/2017.8.JNS163222. Epub 2018 Feb 18. PMID 29451447
- [Background] Quintero JE, Slevin JT, Gurwell JA, McLouth CJ, El Khouli R, Chau MJ, Guduru Z, Gerhardt GA, van Horne CG. Direct delivery of an investigational cell therapy in patients with Parkinson's disease: an interim analysis of feasibility and safety of an open-label study using DBS-Plus clinical trial design. BMJ Neurol Open. 2022 Jul 14;4(2):e000301. doi: 10.1136/bmjno-2022-000301. eCollection 2022. PMID 35949912